CLINICAL TRIAL: NCT05261867
Title: Cardioprotective Effect of Sodium-Glucose Cotransporter-2 Inhibitors (SGLT2-I) in Diabetic Patients With Acute Myocardial Infarction
Brief Title: Cardioprotective Effect of SGLT2-I in Diabetic Patients With AMI (SGLT2-I AMI PROTECT Study)
Acronym: SGLT2-I AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Maggiore Hospital Carlo Alberto Pizzardi (Other); VZW Cardiovascular Research Center Aalst (Other); Cardarelli Hospital (Other); Azienda Ospedaliera Sant'Anna e San Sebastiano (Other); Azienda Ospedaliera "Sant'Andrea" (Other); Alexandrovska University Hospital (Other); Niguarda Hospital (Other); University of Campania Luigi Vanvitelli (Other); ASST Grande Ospedale Metropolitano Niguarda (Other)
Responsible Party: Sponsor
Other Study IDs: SGLT2I001
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus; Acute Coronary Syndrome
Keywords: SGLT2-I; Acute myocardial infarction; Diabetes Mellitus; Prognosis
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients treated with SGLT2-I: Diabetic patients treated with SGLT2-I alone or in combination with other oral anti-diabetic (OAD) agents. Patients were considered in the SGLT2-I group if it was started at least 1 month prior to index hospitalization.
- Diabetic patients treated with other oral anti-diabetic (OAD) agents: Diabetic patients treated with other oral anti-diabetic agents alone.

SUMMARY:
Despite their potential benefits on the heart with pleiotropic mechanisms, the cardioprotective effects of new glucose-lowering SGLT-2 inhibitors in patients with myocardial infarction - both in the acute and chronic phase - have never been explored.

The key point of the project will be the evaluation of the cardioprotective effect and the potential prognostic benefit of SGLT-2 inhibitors in patients with diabetes and acute myocardial infarction.

DETAILED DESCRIPTION:
Classically, the physiopathology of myocardial infarction is linked to the presence of coronary atherosclerosis. According to the European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA) Guidelines of the fourth Universal definition, type 1 myocardial infarction (MI), the most frequent cause was atherothrombotic plaque (the mechanism of plaque erosion, rupture, fissuring with an athero-thrombotic)(1) In acute myocardial infarction, early restoration of epicardial and myocardial blood flow is of paramount importance to limit infarction size and create optimum conditions for favorable long-term outcome. Currently, restoration of epicardial blood flow is preferably and effectively obtained by primary percutaneous coronary intervention (PPCI). After opening the occluded artery, however, the reperfusion process itself causes damage to the myocardium, the so called "reperfusion injury". The phenomenon of reperfusion injury is incompletely understood and currently there is no established therapy for preventing it. Contributory factors are intramyocardial edema with compression of the microvasculature, oxidative stress, calcium overload, mitochondrial transition pore opening, micro embolization, neutrophil plugging and hyper contracture. This results in myocardial stunning, reperfusion arrhythmias and ongoing myocardial necrosis (2,3). There is general agreement that a large part of the cell death caused by myocardial reperfusion injury occurs during the first few minutes of reperfusion, and that early treatment is required to prevent it.

According to current guidelines, drug therapy administrated for acute myocardial infarction includes antiplatelets (against atherosclerotic plaque and stent thrombosis), renin-angiotensin-aldosterone system (RAAS) inhibitors, beta-blockers and lipid-lowering therapy (primarily with statins).

Due to their high efficacy, excellent tolerability, and their ability to reduce major adverse cardiovascular events in large clinical trials, SGLT2 inhibitors have been tested in a variety of preclinical studies and it was demonstrated to reduce acute myocardial ischemia-reperfusion (I/R) injury (4).

Four-week pre-treatment with dapagliflozin could decrease infarct size in rats with obese insulin resistance which underwent cardiac ischemic-reperfusion injury (5) and a recent experimental study demonstrated that acute dapagliflozin administration during cardiac I/R injury exerted cardioprotective effects by attenuating cardiac infarct size, increasing left ventricular function and reducing arrhythmias (6). Moreover, in rats with previous myocardial infarct, dapagliflozin treatment beginning one day after left anterior descending coronary artery ligation could decrease myofibroblast infiltration and myocardial fibrosis (7).

Finally, a preregistered meta-analysis (PROSPERO), that included placebo-controlled, interventional studies of small and large animal models of myocardial ischaemia-reperfusion injury, testing the effect of SGLT2 inhibitor treatment on myocardial infarct size concluded that the glucose-lowering SGLT2 inhibitors reduce myocardial infarct size in animal models independent of diabetes status (8).

Despite its potential benefits on the heart with pleiotropic mechanisms, the cardioprotective effects of new glucose-lowering SGLT-2 inhibitors in patients with myocardial infarction - both in the acute and chronic phase- have never been explored.

The key point of the project will be the evaluation of the cardioprotective effect and the potential prognostic benefit of SGLT-2 inhibitors in patients with diabetes and acute myocardial infarction.

The investigators' findings could provide significant insights for future clinical trials on SGLT-2 inhibitors treatments in patients with ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y old
* STEMI/NSTEMI diagnosed according to ESC guidelines undergoing reperfusion treatment with percutaneous transluminal coronary angioplasty (PTCA).
* Known type II diabetes mellitus treated with oral antidiabetic drugs

Exclusion Criteria:

* Type I diabetes mellitus or type II diabetes mellitus treated only with insulin therapy alone or in combination with other anti-diabetic drugs.
* Patients treated with Coronary artery bypass grafting (CABG) after the coronary angiography (CAG) (NSTEMI)
* Previous CABG
* Severe valvular heart disease.
* Contraindications for secondary medical prevention therapy approved for myocardial infarctions, like beta-blockers, angiotensin-converting enzyme inhibitor(ACEI )/angiotensin receptor blocker (ARBs), antiplatelets, statins. All patients will be treated with optimal secondary prevention therapy suggested by the current ESC guidelines.
* Patients who start SGLT2 therapy after the acute index event.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with STEMI/NSTEMI diagnosed according to ESC guidelines undergoing reperfusion treatment with percutaneous transluminal coronary angioplasty (PTCA) with known type II diabetes mellitus treated with oral antidiabetic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, recurrent AMI, and hospitalization for HF (MACE). | Through study completion, an average of 2 year
  Composite of cardiovascular death, recurrent AMI, and hospitalization for HF (MACE).

SECONDARY OUTCOMES:
Intra-hospital cardiovascular death | Up to 30 days
  Intra-hospital cardiovascular death mortality included deaths that result from an AMI, sudden cardiac death, heart failure, stroke, and other cardiovascular causes during the hospitalization.
Intra-hospital atrial and ventricular arrhythmias | Up to 30 days
  Ventricular arrhythmias were defined as a cardiac arrhythmia of three or more consecutive complexes originating from the ventricles at a rate of greater than 100 beats per minute. We included both sustained (lasting 30 sec or more) and non-sustained (lasting less than 30 sec) ventricular arrhythmias due to similar risk of adverse cardiovascular outcomes associated with both these types.
Reduction of the infarct size | Up to 30 days
  Myocardial infarct size was estimated using high-sensitivity troponin (at the moment of hospital admission and every 3-6 hours thereafter for the following 24 hours) and the left ventricular end-diastolic volume (LVEDV) and the biplane left ventricular ejection fraction (LVEF).
Reduction of the inflammatory response. | Up to 30 days
  The inflammatory response was evaluated using the following parameters: C reactive protein (CRP), white blood cells - leukocytes and neutrophils count, neutrophil to lymphocyte ratio (NLR), neutrophil to platelet ratio (NPR), platelet to lymphocytes ratio (PLR), C-Reactive Protein. In particular, NLR is the ratio of neutrophil and lymphocyte counts, NPR is the ratio of neutrophil and platelet counts, and PLR is obtained by dividing the platelet count by the lymphocytes. Patients with concomitant basal values of CRP and NLR above the median were considered to have an inflammatory response.
Contrast-induced acute kidney injury | Through study completion, an average of 1 year
  Contrast-induced acute kidney injury is defined as an increase in sCr by 0.3 mg/dL or an increase in creatinine to ⩾1.5 times baseline within 3 to 5 days following contrast exposure.
Length of hospital stay | Up to 30 days
  Length of hospitalization (days)
All-cause mortality | Through study completion, an average of 2 year
  All-cause mortality included all causes of death for the population during the follow-up.
Cardiovascular mortality | Through study completion, an average of 2 year.
  Cardiovascular death consisted of deaths that result from an AMI, sudden cardiac death, heart failure, stroke, and other cardiovascular causes.
Heart failure hospitalization. | Through study completion, an average of 2 year.
  Heart failure re-hospitalization was evaluated according to the ESC Guidelines and consisted of unscheduled hospital admission for a primary diagnosis of HF in which the patient presented typical signs, symptoms, and diagnostic testing consistent with the diagnosis of HF and consequently received HF-directed therapy.
Recurrent AMI | Through study completion, an average of 2 year
  Recurrent acute myocardial infarction.
Any coronary revascularization | Through study completion, an average of 2 year
  Clinically indicated target vessel revascularization for significant renarrowing.

CONTACTS AND LOCATIONS:
Locations (7):
- Cardiovascular Center Aalst, OLV-Clinic, Aalst, Belgium, Aalst, Belgium
- Alexandrovska University Hospital, Sofia, Bulgaria, Sofia, Bulgaria
- Italy (5):
  - Policlinico Sant'Orsola, Bologna
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta, Caserta
  - ASST Grande Ospedale Metropolitano Niguarda, Milano, Milan
  - Università Vanvitelli, Ospedale Cardarelli, Napoli, Napoli
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Result] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Result] Andreadou I, Bell RM, Botker HE, Zuurbier CJ. SGLT2 inhibitors reduce infarct size in reperfused ischemic heart and improve cardiac function during ischemic episodes in preclinical models. Biochim Biophys Acta Mol Basis Dis. 2020 Jul 1;1866(7):165770. doi: 10.1016/j.bbadis.2020.165770. Epub 2020 Mar 17. PMID 32194159
- [Result] Tanajak P, Sa-Nguanmoo P, Sivasinprasasn S, Thummasorn S, Siri-Angkul N, Chattipakorn SC, Chattipakorn N. Cardioprotection of dapagliflozin and vildagliptin in rats with cardiac ischemia-reperfusion injury. J Endocrinol. 2018 Feb;236(2):69-84. doi: 10.1530/JOE-17-0457. Epub 2017 Nov 15. PMID 29142025
- [Result] Lahnwong C, Palee S, Apaijai N, Sriwichaiin S, Kerdphoo S, Jaiwongkam T, Chattipakorn SC, Chattipakorn N. Acute dapagliflozin administration exerts cardioprotective effects in rats with cardiac ischemia/reperfusion injury. Cardiovasc Diabetol. 2020 Jun 15;19(1):91. doi: 10.1186/s12933-020-01066-9. PMID 32539724
- [Result] Lee TM, Chang NC, Lin SZ. Dapagliflozin, a selective SGLT2 Inhibitor, attenuated cardiac fibrosis by regulating the macrophage polarization via STAT3 signaling in infarcted rat hearts. Free Radic Biol Med. 2017 Mar;104:298-310. doi: 10.1016/j.freeradbiomed.2017.01.035. Epub 2017 Jan 26. PMID 28132924
- [Result] Sayour AA, Celeng C, Olah A, Ruppert M, Merkely B, Radovits T. Sodium-glucose cotransporter 2 inhibitors reduce myocardial infarct size in preclinical animal models of myocardial ischaemia-reperfusion injury: a meta-analysis. Diabetologia. 2021 Apr;64(4):737-748. doi: 10.1007/s00125-020-05359-2. Epub 2021 Jan 23. PMID 33483761
- [Derived] Paolisso P, Bergamaschi L, Gragnano F, Gallinoro E, Cesaro A, Sardu C, Mileva N, Foa A, Armillotta M, Sansonetti A, Amicone S, Impellizzeri A, Esposito G, Morici N, Andrea OJ, Casella G, Mauro C, Vassilev D, Galie N, Santulli G, Marfella R, Calabro P, Pizzi C, Barbato E. Outcomes in diabetic patients treated with SGLT2-Inhibitors with acute myocardial infarction undergoing PCI: The SGLT2-I AMI PROTECT Registry. Pharmacol Res. 2023 Jan;187:106597. doi: 10.1016/j.phrs.2022.106597. Epub 2022 Dec 5. PMID 36470546
- [Derived] Cesaro A, Gragnano F, Paolisso P, Bergamaschi L, Gallinoro E, Sardu C, Mileva N, Foa A, Armillotta M, Sansonetti A, Amicone S, Impellizzeri A, Esposito G, Morici N, Oreglia JA, Casella G, Mauro C, Vassilev D, Galie N, Santulli G, Pizzi C, Barbato E, Calabro P, Marfella R. In-hospital arrhythmic burden reduction in diabetic patients with acute myocardial infarction treated with SGLT2-inhibitors: Insights from the SGLT2-I AMI PROTECT study. Front Cardiovasc Med. 2022 Sep 27;9:1012220. doi: 10.3389/fcvm.2022.1012220. eCollection 2022. PMID 36237914
- [Derived] Paolisso P, Bergamaschi L, Santulli G, Gallinoro E, Cesaro A, Gragnano F, Sardu C, Mileva N, Foa A, Armillotta M, Sansonetti A, Amicone S, Impellizzeri A, Casella G, Mauro C, Vassilev D, Marfella R, Calabro P, Barbato E, Pizzi C. Infarct size, inflammatory burden, and admission hyperglycemia in diabetic patients with acute myocardial infarction treated with SGLT2-inhibitors: a multicenter international registry. Cardiovasc Diabetol. 2022 May 15;21(1):77. doi: 10.1186/s12933-022-01506-8. PMID 35570280